CLINICAL TRIAL: NCT04819971
Title: Efficacy and Safety of Perioperative Chemotherapy Combined With Tislelizumab and Trastuzumab in Patients With HER2-positive Resectable Gastric or Gastr-oesophageal Junction Carcinoma (GC/EGJ) -- a Prospective, Single-arm, Phase II Study
Brief Title: Study of Perioperative Chemotherapy Combined With Tislelizumab and Trastuzumab in the Treatment of GC/EGC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Feng Wang, Associate Chief Physician, The First Affiliated Hospital of Zhengzhou University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TIS-HER2GC-PERIOPERATIVE-IIT
Record Dates: First submitted 2021-03-21; First posted 2021-03-29 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Stomach Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Trastuzumab; Docetaxel; S 1 (combination); Oxaliplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TTC (Experimental)
  Interventions: Drug: Tirelizumab; Drug: Trastuzumab; Drug: Docetaxel; Drug: S1; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Tirelizumab — tislelizumab (intravenously, 200 mg on day 1 of every cycle for 4 preoperative and 12 postoperative cycles)
Drug: Trastuzumab — Trastuzumab(intravenously, 8 mg/kg loading dose, then 6 mg/kg on days 1 of every cycle for 4 preoperative and 12 postoperative cycles)
Drug: Docetaxel — docetaxel (intravenously, 50 mg/m2 on day 1 of every cycle for 3 preoperative cycles)
Drug: S1 — S1 (orally, 400mg/m2 BID on day 1~14 of every cycle for 3 preoperative and 3 postoperative cycles )
Drug: Oxaliplatin — Oxaliplatin(intravenously, 100 mg /m2 on day 1 of every cycle for 3 preoperative cycles ;130mg /m2 on day 1 of every cycle for 3 postoperative cycles.

SUMMARY:
Perioperative chemotherapy improves overall survival (OS) and disease-free survival (DFS) compared with surgery alone in patients with resectable gastric adenocarcinoma (GA) or gastro-oesophageal junction adenocarcinoma (GEJA). The addition of tislelizumab and trastuzumab to chemotherapy improves outcomes in patients with HER2-positive advanced gastric cancer (GC), and the investigators aimed to explore its role in the perioperative setting.

DETAILED DESCRIPTION:
This study will evaluate the pathologic complete response rate of a perioperative chemotherapy combined with tislelizumab and Trastuzumab in patients with resectable gastric cancer. Prior to surgery to resect the tumor, tislelizumab (intravenously, 200 mg on day 1 of every cycle) and trastuzumab (intravenously, 8 mg/kg loading dose, then 6 mg/kg on days 1 of every cycle) will be administered for four cycles and the perioperative chemotherapy contains docetaxel (intravenously, 50 mg/m2 on day 1 of every cycle) and S1 (orally, 400mg/m2 BID on day 1~14 of every cycle) and Oxaliplatin(intravenously, 100 mg /m2 on day 1 of every cycle) will be administered for three cycles prior to surgery.If complete resection, R0 or microscopic residual tumor R1 is achieved, patients will continue with three cycles of SOX and tislelizumab and trastuzumab and then for completion of 12 months treatment with tislelizumab and trastuzumab alone.

ELIGIBILITY:
Key Inclusion Criteria:

* provide archive tumor tissue samples or accept fresh tumor tissue biopsy(Sample requirements are: formalin-fixed and paraffin-embedded wax blocks of tumor tissue or at least 20 unstained tumor specimen slides).
* assessed by the surgery can be removed, histology/confirmed HER2 positive cytology and the integration of a stomach esophagus carcinoma.

  * CT2-4CN any C M0 or T any CN +M0, AJCC/UICC TNM staging of gastric cancer (8th edition).
  * The HER2 receptor protein status was assessed by immunohistochemistry (IHC) and fluorescence in situ hybridization (FISH) using the following methods.Tumors with an IHC 3+ score are considered HER2-positive.Patients with immunohistochemical 2+ tumors were given FISH tests to determine FISH positive samples.
  * Abdominal computed tomography (CT), abdominal, pelvic, and/or echo-endoscopy were performed 2 weeks before surgery to assess resectability.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 or 2.
* have no received no any anti-tumor treatment, including surgery, chemotherapy, targeted therapy, immune therapy.
* Adequate organ function (No blood transfusion or hematopoietic stimulating factor therapy was received within 14 days. Absolute neutrophil count (ANC) ≥1.5×109/L Platelet count ≥75×109/L Hemoglobin ≥80 g/L. Serum total bilirubin ≤1.5×ULN. total bilirubin must be <3×ULN) Prothrombin time/international normalized ratio (PT/INR) ≤1.5×ULN and activated partial thromboplastin time (aPTT) ≤1.5×ULN.Aspartate transaminase (AST) and alanine aminotransferase (ALT) ≤3×ULN. For subjects with liver metastases, AST and ALT must be ≤5×ULN for subjects with liver metastases. Creatinine clearance rate (Ccr) ≥50ml/min（according to the Cockcroft-Gault formula）. Urine protein qualitative≤1+ ;Or urinary protein qualitative ≥2+, 24 hours urinary protein < 1g)

Key Exclusion Criteria:

* A history of any other malignancy in the past 5 years (except carcinoma in situ or basal cell carcinoma of the skin or squamous cell carcinoma of the skin)
* Received other unmarketed investigational drug or therapy within 4 weeks prior to initial investigational drug use.
* A major organ surgery (excluding needle biopsy) or significant trauma occurred within 4 weeks prior to initial investigational drug use.
* Requires systemic treatment with either corticosteroids (>10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration to treat a current condition.

Exceptions include: topical, ocular, intraarticular, intranasal, and inhaled glucocorticoids;Short-term use of glucocorticoids for preventive treatment (e.g. to prevent contrast allergy)

* Use of immunoregulatory drugs, including but not limited to thymosin, interleukin-2, interferon, etc., within 14 days prior to initial use of the study drug.
* Has been administered a live vaccine within 4 weeks prior to Cycle1 Day 1.
* Previous recipient of allogeneic hematopoietic stem cell transplantation or organ transplantation.
* Previous adverse reactions to other medications have not recovered to CTCAE 5.0 level ≤1 (Other toxicities, such as hair loss, were not considered to pose a safety risk).
* Symptomatic peripheral neuropathy was evaluated as > 2 with CTCAE 5.0.
* Has central nervous system metastases or meningeal metastases.
* Inability to swallow medications orally, or other gastrointestinal diseases (such as total intestinal obstruction, etc.) that may affect the absorption of oral medications.
* Patients who had an active infection within 1 week prior to the first use of the study drug and who currently require systemic anti-infective therapy.
* has a history of alcohol or drug abuse or dependence.
* Known history of Human Immunodeficiency Virus (HIV).
* Untreated chronic hepatitis B viral (HBV) infection or chronic HBV carrier with HBV DNA ≥200 IU/mL (or 1000 copies/mL),prophylaxis antiviral therapy other than interferon is allowed ,or active hepatitis C virus (HCV) should be excluded.
* Current patients with interstitial lung disease.
* Has a history of severe cardiovascular and cerebrovascular disease, including but not limited to: has serious heart rhythm or abnormal conduction;Acute coronary syndrome, congestive heart failure, aortic dissection, stroke, or other grade 3 or higher cardiovascular and cerebrovascular events occurred within 6 months prior to D1 ;New York heart association (NYHA), cardiac function class II or higher and left ventricular ejection fraction (LVEF) < 50%; clinical uncontrol of high blood pressure.
* Patients with active, or previous and recurrent autoimmune diseases (such as systemic lupus erythematosus, rheumatoid arthritis, vasculitis, etc.) were excluded from patients with clinically stable autoimmune thyroid disease.
* Grade 3 or higher arteriovenous thromboembolism events or bleeding events occurred within 6 months prior to the first use of the study drug;Or present with grade ≥2 bleeding or factors determined by the investigator to have a higher blood risk (such as active gastrointestinal ulcer or esophageal varicose veins or tumor invasion of major blood vessels).
* Gastrointestinal perforation, abdominal fistula or intraperitoneal abscess occurred within 6 months prior to the first use of the study drug;Or a risk factor for cavity perforation/fistula formation (e.g., tumor infiltration of the outer wall of the cavity wall) currently identified by the investigator.
* Patients who allergies to the study drugs.
* People with mental disorders or poor compliance.
* Women who are pregnant or lactating.
* The investigator considers the subject to have a history of other serious systemic disease or for other reasons unsuitable for participation in this clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With Pathological Complete Response (pCR) | 2 years
  pCR was defined as an absence of any invasive cancer cell of the primary tumor after the time of major neoadjuvant chemotherapy, with or without surgery.

SECONDARY OUTCOMES:
Percentage of Participants With Complete Tumor Resection (R0) | 75 days
  R0 resection was defined as having performed a complete resection of the tumor with adequate tumor-free margins and regional lymph node extirpation.
Percentage of Participants With Disease-free Survival (DFS) | 2 years
  DFS was the time elapsed from the time of surgery (for complete resection [R0] participants) until the date on which progression or death from any cause was documented (whichever occured first). Progression was defined as target lesions greater than (>) 20 percent (%) increase in the sum of the longest diameter (SLD) taking as reference the smallest SLD recorded since the treatment started (nadir) and minimum 5 millimeter (mm) increase over the nadir. When the sum becomes very small, increases within the measurement error (2-3 mm) can lead to a 20% increase. Participants who did not present progression and who had not died were censored on the last date on which it was known that there was no progression (last response assessment).
Overall Survival (OS) | 2 years
  OS was defined as the time from randomization to death due to any cause. Participants without documented death at the time of the final analysis were censored at the date of the last follow-up. OS was analyzed using the Kaplan-Meier method and median OS (95% CI) in months was reported for PD-L1 positive participants by treatment group.
Percentage of All Participants That Discontinued Study Treatment Due to AE | 2 years
  An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE could therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a pre-existing condition that was temporally associated with the use of the Sponsor's product was also an AE. The percentage of participants that discontinued study treatment due to an AE was reported for all participants by treatment group.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China